CLINICAL TRIAL: NCT05324475
Title: Maintaining Immune and Mitochondrial Functions in Old Adults With SAfe Nutrition: the MIMOSA Study.
Brief Title: Maintaining Immune and Mitochondrial Functions in Old Adults With SAfe Nutrition.
Acronym: MIMOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patrizia D'Amelio (Other)
Responsible Party: Sponsor-Investigator, Patrizia D'Amelio, associated professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIMOSA
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malnutrition; Sarcopenia
Keywords: malnutrition; sarcopenia; immune system; Mitochondria; oxydative stress; inflammaegeing; branch-chained aminoacids; micronutrients; nutrition
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Intervention Model Description: three arms study double blind placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention nutrients will be delivered as powder in sachets identified as B (BCAA, 4 gr) or C (mixture of micronutrients, 4 gr), placebo sachets identified as A will contain maltodextrin, (4 gr); the sachets will be mixed by the patients in a juice. Blinding will be maintained until interim evaluation and after for the full trial. In order to assure the blinding the sachets will be opaque identified by a single letter ready to be mixture with a juice with similar taste and texture between the different formulations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (SC) (Placebo Comparator): nutritional counselling (SC) + Placebo: These patients will receive Oral Nutrient Supplementation (ONS) and maltodextrin 4 g
  Interventions: Dietary Supplement: standard treatment + placebo
- Branch-chained aminoacids (Experimental): In addition to the ONS these patients will receive 4 gram per day of BCAAs mixture. Ratio between the BCAAs will be Leucine/Isoleucine/Valine=2:1:1.
  Interventions: Dietary Supplement: BCAA
- Micronutrients (Experimental): In addition to the ONS the patients will receive a combination of micronutrients and PUFA
  Interventions: Dietary Supplement: Micronutriments

INTERVENTIONS:
Dietary Supplement: BCAA — daily administration of oral nutritional supplements (ONS) 1) providing whole proteins together with dietary advice according with the ESPEN nutrition guidelines. All the patients will receive the standard commercially available product used at CHUV (Resource protein ®, nestle) and nutritional counselling (SC) and 4 gram per day of BCAAs mixture. Ratio between the BCAAs will be Leucine/Isoleucine/Valine=2:1:1
  Arms: Branch-chained aminoacids
Dietary Supplement: Micronutriments — daily administration of oral nutritional supplements (ONS) 1) providing whole proteins together with dietary advice according with the ESPEN nutrition guidelines. All the patients will receive the standard commercially available product used at CHUV (Resource protein ®, nestle ) and nutritional counselling (SC) and Vitamin A 1200 mg RE, Vitamin D3 2000 IU, Thiamine B1 100 mg, Cobalamin B12 10 mcg, Ascorbic acid C 200 mg, Iron 30 mg, Selenium 100 mcg, Zinc 20 mg, Omega-3 PUFA 1 g
  Arms: Micronutrients
Dietary Supplement: standard treatment + placebo — daily administration of oral nutritional supplements (ONS) 1) providing whole proteins together with dietary advice according with the ESPEN nutrition guidelines. All the patients will receive the standard commercially available product used at CHUV (Resource protein ®, nestle ) and nutritional counselling (SC) and maltodextrin 4 g as placebo
  Arms: Standard treatment (SC)

SUMMARY:
Aging is associated with an increased inflammation named "inflammageing" and with an altered immune response. Different mechanisms have been proposed to explain the phenomenon of inflammageing and increased oxidative stress: deficiencies in essential amino acids, and some micronutrients have an important impact and may induce immune cell dysregulation. Mitochondrial dysfunction may explain the complex relationship between malnutrition sarcopenia, immune dysfunction and aging.

Therefore, a personalized nutritional strategy aiming to improve mitochondrial function, decrease oxidative stress, down-regulate inflammation and restore immunity appears to be a logical approach in order to treat malnutrition and its biological and clinical consequences.

MIMOSA will investigate the role of nutritional supplements in rescuing altered mitochondrial function and redox state imbalance.

DETAILED DESCRIPTION:
The study participants will all receive optimal standard care ensuring the optimal protein and energy intakes, with at least 1 g protein per kg body weight and day, and 30 kcal per kg body weight and day (or the measured energy expenditure (EE) value). This will be realized by the daily administration of oral nutritional supplements (ONS) providing whole proteins together with dietary advice [according with the ESPEN nutrition guidelines. All the patients will receive the standard commercially available product used at CHUV (Resource protein ®, Nestlé) and nutritional counselling (SC).

All participants included in this study will receive daily, the oral nutritional supplement (ONS), one sachet and two capsule (for blinding purpose).

The intervention nutrients will be delivered as follows:

* BCAA: 1 sachet containing 4 g of BCAA (details in Table 1)
* Micronutrients: 1 sachet containing 4 g of the micronutrient blend and 2 capsules containing 0.6 g of OMEGA 3 PUFA (details in table 1).

The placebos will be delivered like this:

-1 sachet containing 1 g of maltodextrin and 2 capsules containing 0.6 g of coconut oil. (detailed in Table 1).

The duration of the intervention will be 6 weeks, but at least 4 weeks After enrollment patients will be subjected to evaluation of muscle mass by bioimpedance (BIA), muscle strength will be by handgrip strength and muscle performance by the Short Performance Physical Battery (SPPB).

Nutritional status will be evaluated by the Mini Nutritional Assessment short form (MNA-SF), Nutrition Risk screening (NRS) score and Body mass index (BMI). Energy expenditure (EE) will be measured by indirect calorimetry using a canopy.

Moreover appropriate experiments will be carried out in order to evaluate mitochondrial bioenergetics, replication, and fusion, as well as of redox state.

Analyses of inflammageing and immune-senescence will be done by appropriate lab experiments.

Micronutrient status will be measured by ELISA or HPLC and ICPMS respectively. Patients will be evaluated at inclusion, at rehabilitation discharge, and one and two months after rehabilitation discharge. The volume of blood required for the above investigations will be 3 x 30 ml over the 2-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75 years
* Patients entering a rehabilitation program
* Diagnosis of malnutrition defined by a MNA-SF (mini-nutritional assessment short form) score below 11 points.
* Commitment to accept the nutritional supplement proposed, willing and able to give written informed consent
* Ability to understand and comply with the requirements of the study

Exclusion Criteria:

* Presence of malignancy,
* Life expectancy of less than two months calculated by Multidimensional Prognostic Index (MPI ),
* Congestive heart failure (NYHA IV),
* Chronic renal disease (creatinine clearance <40 ml/min calculated by cockroft),
* Liver cirrhosis (Child B-C),
* Tube/percutaneous endoscopic gastrostomy feeding or parenteral nutrition,
* Severe dysphagia,
* Mini-Mental State Examination (MMSE)≤18 and MNA>11 points. MMSE ≥ 18 identifies patients with mild form of cognitive impairment; those patients generally do not have problems in swallowing and are able to take drugs.
* Severe anaemia (Hb<10 g/l) or leukopenia (<2G/l).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial ATP production (nmol/ml) | change vesus baseline at 30, 60 days after discharge
  Production of ATP will be measured using the ATP Bioluminescent Assay Kit
Change in redox state (plasmatic concentration of metabolites) | change vesus baseline at 30, 60 days after discharge
  analyses of thiometabolome contains: methionine, methionine sulfone, methionine sulfoxide, cysteine, homocysteine, homocystine, cystathionine, formylmethionine, cystine, glutathione, glutathione disulfide, taurine, S-adenosylmethionine, S-adenosylhomocysteine, N-acetylcysteine, cysteic acid, serine, glycine, glutamic acid, lypoic acid, selenocysteine, thioctic acid, pyruvic acid.
Change in mitochondrial electron flux (nmol cit/min/mg prot) | change vesus baseline at 30, 60 days after discharge
  The activity of Complex I and III will be measured on non-sonicated mitochondrial samples

SECONDARY OUTCOMES:
change micronutrients status (concentration of micronutrients) | change versus baseline at 60 days after discharge
  Blood levels of Vitamins A, B12, D and E, as well as of trace elements Cu, Fe, Se, and Zn will be determined by ELISA or HPLC and ICPMS
change in inflammation | change versus baseline at 30, 60 days after discharge
  Production of pro-inflammatory cytokines involved in inflammageing and in muscle waste will be measured by ELISA technique; we will measure IL-6 and TNF-alpha (pg/ml).
change phase angle (score) | change versus baseline at rehab discarge (21 days), 30, 60 days after discharge
  Bioelectrical impedance analysis (BIA) will be carried out
muscle function (score) | change versus baseline at rehab discarge (21 days), 30, 60 days after discharge
  Short performance physical battery will be used to measure muscle performance
muscle mass (Kg/body weight) | change versus baseline at rehab discarge (21 days), 30, 60 days after discharge
  Bioelectrical impedance analysis (BIA) will be used to measure muscle mass
muscle strength (Kg) | change versus baseline at rehab discarge (21 days), 30, 60 days after discharge
  Hand grip will be used to measure muscle strenght
change in perceived health status (score) | change versus baseline at rehab discarge (21 days), 30, 60 days after discharge
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia D'amelio, Principal Investigator — Service de gériatrie et réadaptation gériatrique-CHUV
Locations (1):
- CHUV, Lausanne, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared according to the F.A.I.R. principles as follows. Findable- Accessible. All data collected will be uploaded to the Redcap research data repository after anonymization.
  Interoperable. The majority of the raw data produced will be in standard formats for which there is suitable open source software available.
  Reusable. Data publicly available will use the Creative Commons Attribution version 3.0 (http://creativecommons.org/licenses/by/3.0/) license that permits free sharing and adaptation of the licensed data with the restrictions depicted above and any related scientific publications as well as documenting any changes. Each dataset will contain appropriate citation details in the accompanying README file.
  We will make data open immediately if not sensitive for IP protection. Data with sensitive IP will be made available after 5 years from the end of the project,
Supporting Information: Study Protocol, ICF, CSR
Time Frame: We will make data open immediately if not sensitive for IP protection. Data with sensitive IP will be made available after 5 years from the end of the project
Access Criteria: upon reasonable request to the PI